CLINICAL TRIAL: NCT01178099
Title: A Pharmacokinetic and Pharmacodynamic Assessment of Prasugrel in Healthy Adults and Adults With Sickle Cell Disease
Brief Title: An Assessment of Prasugrel on Healthy Adults and Sickle Cell Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13746; H7T-MC-TAEJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Results first posted 2012-02-15 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-01

CONDITIONS: Anemia, Sickle Cell
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prasugrel (Experimental): Participants received a single 10 milligram (mg) dose on Day 1 (single dose [SD]), followed by either 5 mg/day (for participants<60 kilograms [kg]) or 7.5 mg/day (for participants≥60 kg) for an additional 11 days (multiple dose [MD]).
  Interventions: Drug: Prasugrel

INTERVENTIONS:
Drug: Prasugrel — Oral, daily for 12 days
  Other Names: LY650315; CS747; Effient; Efient

SUMMARY:
The purpose of this study is to measure the exposure to prasugrel's active metabolite and the pharmacodynamic effects of prasugrel treatment in people with Sickle Cell Disease (SCD).

ELIGIBILITY:
Inclusion Criteria:

* Are 50 to 100 kilograms (kg), inclusive, at the time of screening.
* Have signed informed consent.
* If female, agree to use a reliable method of birth control during the study or are women not of child-bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause.
* Control Subjects - Are healthy adults as determined by medical history, physical examination, and other screening procedures.
* Sickle cell disease (SCD) Subjects - Subjects on hydroxyurea must be on a stable dose for the 30 days prior to enrollment without signs of hematologic toxicity at screening.
* SCD Subjects - Are adults with SCD (hemoglobin SS [HbSS], Hb S beta0 thalassemia, Hb SC or Hb S beta+ thalassemia genotype) without a diagnosis of acute vaso-occlusive crisis (VOC) requiring medical intervention in an emergency department, infusion center, or as an inpatient) within the month prior to screening.

Exclusion Criteria:

* Have a concomitant medical illness (for example, terminal malignancy) that, in the opinion of the investigator, is associated with reduced survival over the expected treatment period (approximately 1 month).
* Exhibit severe hepatic dysfunction (cirrhosis, portal hypertension, or alanine aminotransferase [ALT] for aspartate aminotransaminase [AST]≥3 times upper limit of normal [ULN]).
* Exhibit severe renal dysfunction defined as Cockcroft-Gault creatinine clearance<30 milliliters per minute (ml/min), or requiring chronic dialysis. Creatine clearance = [(140-Age) * Mass (in kg)] \ [72 * Serum creatinine (in milligrams per deciliter [mg/dL])].
* Exhibit any contraindication for antiplatelet therapy.
* Have a history of intolerance or allergy to approved thienopyridines.
* Exhibit any signs or symptoms of an infection.
* Have a hematocrit <18%.
* Exhibit any history of bleeding diathesis, bleeding requiring in-hospital treatment, or papillary necrosis.
* Have active internal bleeding.
* Have a history of spontaneous bleeding requiring in-hospital treatment.
* Have gross hematuria or >300 red blood cells (RBC)/high-powered field (HPF) on urinalysis at the time of screening.
* History of previous intraocular hemorrhage which required treatment with surgery or laser, or evidence of active intraocular haemorrhage.
* Have a prior history of transient ischemic attack (TIA), ischemic stroke, hemorrhagic stroke or other intracranial hemorrhage.
* Have a known history of intracranial neoplasm, arteriovenous malformation, or aneurysm.
* Have clinical findings, in the judgment of the investigator, associated with an increased risk of bleeding.
* Have an international normalized ratio (INR) known to be >1.5 (INR testing not required for study entry).
* Have had recent surgery (within 30 days prior to screening) or are scheduled to undergo surgery within the next 60 days.
* Have a recent history of clinically significant menorrhagia.
* Have used any aspirin, warfarin, or thienopyridine in the 10 days prior to enrollment.
* Have used any non-aspirin non-steroidal anti-inflammatory drug (NSAID) in the 3 days prior to enrollment.
* Anticipate using aspirin, warfarin, NSAID, thienopyridine or other antiplatelet agent during the study period.
* Are women who are known to be pregnant, who have given birth within the past 90 days, or who are breastfeeding.
* Regular use of drugs of abuse and/or unacceptable positive findings on urinary drug screening (a positive urinary drug screening for sleep inducers or pain medications in subjects with SCD will be considered as an acceptable finding).
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device or off-label use of a drug or device, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317 615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, UK, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Prasugrel Healthy Participants: Participants received a single 10-milligram (mg) dose on Day 1 (single dose [SD]), followed by either 5 mg/day (for participants<60 kilograms [kg]) or 7.5 mg/day (for participants≥60 kg) for an additional 11 days (multiple dose [MD]).
- Prasugrel Sickle Cell Disease: Participants received a single 10-mg dose on Day 1 (SD), followed by either 5 mg/day (for participants<60 kg) or 7.5 mg/day (for participants≥60 kg) for an additional 11 days (MD).
Period: Overall Study
Arm/Group | Prasugrel Healthy Participants | Prasugrel Sickle Cell Disease
Started | 13 | 13
Completed | 13 | 12
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Prasugrel 10 mg SD; 5 mg MD (Healthy): Participants received a single 10-milligram (mg) dose on Day 1 (single dose [SD]), followed by 5 mg/day (for participants<60 kilograms [kg]) for an additional 11 days (multiple dose [MD]).
- Prasugrel 10 mg SD; 7.5 mg MD (Healthy); Prasugrel 10 mg SD; 7.5 mg MD (Sickle Cell Disease): Participants received a single 10-mg dose on Day 1 (SD), followed by 7.5 mg/day (for participants≥60 kg) for an additional 11 days (MD).
- Prasugrel 10 mg SD; 5 mg MD (Sickle Cell Disease): Participants received a single 10-mg dose on Day 1 (SD), followed by 5 mg/day (for participants<60 kilograms [kg]) for an additional 11 days (MD).
- Total: Total of all reporting groups
Arm/Group | Prasugrel 10 mg SD; 5 mg MD (Healthy) | Prasugrel 10 mg SD; 7.5 mg MD (Healthy) | Prasugrel 10 mg SD; 5 mg MD (Sickle Cell Disease) | Prasugrel 10 mg SD; 7.5 mg MD (Sickle Cell Disease) | Total
Number analyzed (Participants) | 4 | 9 | 4 | 9 | 26
Age Continuous [Mean (Standard Deviation); unit: years] | 24.8 (3.0) | 27.6 (6.5) | 28.0 (14.8) | 29.6 (6.8) | 27.9 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 2 | 11
  Male | 0 | 7 | 1 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 3 | 8 | 4 | 9 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 4 | 9 | 16
  White | 1 | 8 | 0 | 0 | 9
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 4 | 9 | 4 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) From Time of Dosing Through the Sampling Time of the Last Quantifiable Concentration [AUC(0-tlast)] for Prasugrel's Active Metabolite, R-138727
Description: The AUC of Prasugrel's active metabolite, R-138727, was calculated through the sampling time of the last quantifiable plasma concentration [AUC(0-tlast)]. Geometric Least Squares (LS) Means were obtained. The log-transformed AUC was analyzed with a mixed effect model with dose, population, dose*population interaction as fixed effects, and participant as a random effect.
Time Frame: Time of dosing up to 8 hours post-dose on Day 1 and Day 12
Population: All participants who received at least 1 dose of the study drug and have evaluable data, excluding participants with an adverse event (AE) of vomiting that occurred at or before 4-hours postdose.
Measure: Least Squares Mean (95% Confidence Interval); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Prasugrel Healthy Participants | Prasugrel Sickle Cell Disease
Number analyzed (Participants) | 13 | 12
nanogram*hour per milliliter (ng*h/mL)
  10 mg SD (overall) | 68.2 [57.9 to 80.5] | 71.5 [60.5 to 84.6]
  7.5 mg MD (N=9, 8) | 50.4 [42.0 to 60.5] | 45.2 [37.2 to 54.8]
  5 mg MD (N=4, 4) | 39.8 [30.3 to 52.3] | 36.0 [27.4 to 47.4]
Statistical Analysis 1: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(AUC) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 1.05, 90% CI 2-sided [0.829 to 1.33] — This is the estimated value for the 10 mg SD (overall)
Statistical Analysis 2: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(AUC) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 0.895, 90% CI 2-sided [0.718 to 1.12] — This is the estimated value for the 7.5 mg MD
Statistical Analysis 3: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(AUC) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 0.905, 90% CI 2-sided [0.656 to 1.25] — This is the estimated value for the 5 mg MD

2. Primary Outcome: Maximum Concentration (Cmax) of Prasugrel's Active Metabolite, R-138727
Description: Cmax was observed from the data and used to calculate Geometric Least Squares (LS) Means. The log-transformed Cmax was analyzed with a mixed effect model with dose, population, dose*population interaction as fixed effects, and participant as a random effect.
Time Frame: Day 1, Day 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: nanogram per milliliter (ng/mL)
Arm/Group | Prasugrel Healthy Participants | Prasugrel Sickle Cell Disease
Number analyzed (Participants) | 13 | 12
nanogram per milliliter (ng/mL)
  10 mg SD (overall) | 67.9 [52.8 to 87.4] | 64.7 [50.1 to 83.7]
  7.5 mg MD (N=9, 8) | 62.5 [47.2 to 82.7] | 38.2 [28.4 to 51.5]
  5 mg MD (N=4, 4) | 40.9 [26.9 to 62.3] | 42.0 [27.6 to 63.9]
Statistical Analysis 1: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(Cmax) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 0.953, 90% CI 2-sided [0.664 to 1.37] — This is the estimated value for the 10 mg SD (overall)
Statistical Analysis 2: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(Cmax) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 0.612, 90% CI 2-sided [0.436 to 0.860] — This is the estimated value for the 7.5 mg MD
Statistical Analysis 3: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(Cmax) = Participant + Population + Dose + Population*Dose + Random Error; Geometric LS Means, SCD:Healthy = 1.03, 90% CI 2-sided [0.625 to 1.68] — This is the estimated value for 5 mg MD

3. Secondary Outcome: Change From Baseline in the Maximum Platelet Aggregation (MPA) to 5 Micromolar (µM) Adenosine Diphosphate (ADP) at Day 12
Description: MPA to 5 μM ADP was assessed by light transmission aggregometry (LTA), an assay that measures platelet aggregation by determining the amount of light transmitted through a cuvette containing the platelet-rich plasma stimulated with a platelet activator, such as ADP, relative to platelet-poor plasma (100% light transmittance). The LTA results were collected as MPA, for which low values indicate strong platelet inhibition.
Time Frame: Baseline, Day 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent aggregation
Arm/Group | Prasugrel Healthy Participants | Prasugrel Sickle Cell Disease
Number analyzed (Participants) | 13 | 11
percent aggregation
  Baseline (Day 1) | 80.4 (23.2) | 73.1 (14.4)
  Change from Baseline at Day 12 (N=12, 7) | -49.9 (18.7) | -33.4 (30.0)
Statistical Analysis 1: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; p = 0.070, ANCOVA — The p-value is from model: Change from Baseline = Baseline + Treatment + Population + Treatment*Population + Random Error

4. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) From Time of Dosing Through the Sampling Time of the Last Quantifiable Concentration [AUC(0-tlast)] of Prasugrel's Inactive Metabolites, R-95913, R-106583, and R-119251
Description: AUC was calculated through the sampling time of the last quantifiable plasma concentration [AUC(0-tlast)]. Geometric Least Squares (LS) Means were obtained. The log-transformed AUC was analyzed with a mixed effect model with dose, population, dose*population interaction as fixed effects, and participant as a random effect.
Time Frame: Day 1, Day 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Prasugrel Healthy Participants | Prasugrel Sickle Cell Disease
Number analyzed (Participants) | 13 | 12
nanogram*hour per milliliter (ng*h/mL)
  10 mg SD (overall) for R-95913 | 52.8 [42.1 to 66.1] | 80.2 [63.8 to 101]
  7.5 mg MD for R-95913 (N=9, 8) | 49.4 [38.5 to 63.4] | 70.9 [54.4 to 92.4]
  5 mg MD for R-95913 (N=4, 4) | 33.6 [23.1 to 48.9] | 47.9 [32.9 to 92.4]
  10 mg SD (overall) for R-106583 | 248 [206 to 300] | 241 [199 to 292]
  7.5 mg MD for R-106583 (N=9, 8) | 213 [173 to 263] | 174 [139 to 217]
  5 mg MD for R-106583 (N=4, 4) | 151 [110 to 207] | 144 [105 to 197]
  10 mg SD (overall) for R-119251 | 32.7 [25.8 to 41.6] | 38.3 [30.1 to 48.9]
  7.5 mg MD for R-119251 (N=9, 8) | 22.2 [17.1 to 29.0] | 23.8 [18.0 to 31.6]
  5 mg MD for R-119251 (N=4, 4) | 20.1 [13.5 to 29.9] | 16.3 [11.0 to 24.3]
Statistical Analysis 1: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(AUC) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 1.52, 90% CI 2-sided [1.10 to 2.10] — This is the estimated value for 10 mg SD (overall) for the R-95913 metabolite
Statistical Analysis 2: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(AUC) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 1.44, 90% CI 2-sided [1.06 to 1.94] — This is the estimated value for 7.5 mg MD for the R-95913 metabolite
Statistical Analysis 3: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(AUC) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 1.43, 90% CI 2-sided [0.918 to 2.21] — This is the estimated value for 5 mg MD for the R-95913 metabolite
Statistical Analysis 4: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(AUC) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 0.971, 90% CI 2-sided [0.742 to 1.27] — This is the estimated value for the 10 mg SD (overall) for the R-106583 metabolite
Statistical Analysis 5: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(AUC) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 0.815, 90% CI 2-sided [0.633 to 1.05] — This is the estimated value for the 7.5 mg MD for the R-106583 metabolite
Statistical Analysis 6: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(AUC) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 0.952, 90% CI 2-sided [0.658 to 1.38] — This is the estimated value for the 5 mg MD for the R-106583 metabolite
Statistical Analysis 7: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(AUC) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 1.17, 90% CI 2-sided [0.833 to 1.65] — This is the estimated value for 10 mg SD (overall) for the R-119251 metabolite
Statistical Analysis 8: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(AUC) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 1.07, 90% CI 2-sided [0.779 to 1.48] — This is the estimated value for 7.5 mg MD for the R-119251 metabolite
Statistical Analysis 9: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(AUC) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 0.813, 95% CI 2-sided [0.510 to 1.30] — This is the estimated value for 5 mg MD for the R-119251 metabolite

5. Secondary Outcome: Change From Baseline in the Residual Platelet Aggregation (RPA) to 5 Micromolar (µM) Adenosine Diphosphate (ADP) at Day 12
Description: RPA is the percentage aggregation as measured by LTA at 6 minutes after the addition of 5 μM ADP. LTA is an assay that measures platelet aggregation by determining the amount of light transmitted through a cuvette containing the platelet-rich plasma stimulated with a platelet activator, such as ADP, relative to platelet-poor plasma (100% light transmittance).
Time Frame: Baseline, Day 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent aggregation
Arm/Group | Prasugrel Healthy Participants | Prasugrel Sickle Cell Disease
Number analyzed (Participants) | 13 | 11
percent aggregation
  Baseline (Day 1) | 76.9 (29.1) | 72.2 (14.1)
  Change from Baseline at Day 12 (N=12, 7) | -70.3 (27.4) | -47.3 (35.6)
Statistical Analysis 1: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; p = 0.018, ANCOVA — [p-value comment as in outcome 3, analysis 1]

6. Secondary Outcome: Inhibition of Platelet Aggregation (IPA) to 5 Micromolar (µM) Adenosine Diphosphate (ADP) at Day 12
Description: IPA is calculated as a percent decrease of maximum platelet aggregation (MPA) from baseline using the following formula:
  ([MPA at baseline - MPA postbaseline] / MPA at baseline) x 100%
Time Frame: Day 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent inhibition
Arm/Group | Prasugrel Healthy Participants | Prasugrel Sickle Cell Disease
Number analyzed (Participants) | 12 | 7
percent inhibition | 61.2 (13.1) | 41.7 (47.3)
Statistical Analysis 1: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; p = 0.060, ANCOVA — [p-value comment as in outcome 3, analysis 1]

7. Secondary Outcome: Change From Baseline in the Maximum Platelet Aggregation (MPA) to 20 Micromolar (µM) Adenosine Diphosphate (ADP) at Day 12
Description: MPA to 20 μM ADP was assessed by light transmission aggregometry (LTA), an assay that measures platelet aggregation by determining the amount of light transmitted through a cuvette containing the platelet-rich plasma stimulated with a platelet activator, such as ADP, relative to platelet-poor plasma (100% light transmittance). The LTA results were collected as MPA, for which low values indicate strong platelet inhibition.
Time Frame: Baseline, Day 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent aggregation
Arm/Group | Prasugrel Healthy Participants | Prasugrel Sickle Cell Disease
Number analyzed (Participants) | 13 | 11
percent aggregation
  Baseline (Day 1) | 85.0 (15.9) | 73.4 (12.9)
  Change from Baseline at Day 12 (N=12, 9) | -43.3 (11.7) | -30.9 (22.6)
Statistical Analysis 1: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; p = 0.219, ANCOVA — [p-value comment as in outcome 3, analysis 1]

8. Secondary Outcome: Change From Baseline in the Residual Platelet Aggregation (RPA) to 20 Micromolar (µM) Adenosine Diphosphate (ADP) at Day 12
Description: RPA is the percentage aggregation as measured by light transmission aggregometry (LTA) at 6 minutes after the addition of 20 μM ADP. LTA is an assay that measures platelet aggregation by determining the amount of light transmitted through a cuvette containing the platelet-rich plasma stimulated with a platelet activator, such as ADP, relative to platelet-poor plasma (100% light transmittance).
Time Frame: Baseline, Day 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent aggregation
Arm/Group | Prasugrel Healthy Participants | Prasugrel Sickle Cell Disease
Number analyzed (Participants) | 13 | 11
percent aggregation
  Baseline (Day 1) | 84.1 (16.7) | 72.2 (12.4)
  Change from Baseline at Day 12 (N=12, 8) | -67.0 (18.1) | -45.5 (32.7)
Statistical Analysis 1: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; p = 0.177, ANCOVA — [p-value comment as in outcome 3, analysis 1]

9. Secondary Outcome: Inhibition of Platelet Aggregation (IPA) to 20 Micromolar (µM) Adenosine Diphosphate (ADP) at Day 12
Description: as for outcome 6
Time Frame: Day 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent inhibition
Arm/Group | Prasugrel Healthy Participants | Prasugrel Sickle Cell Disease
Number analyzed (Participants) | 12 | 9
percent inhibition | 52.6 (13.5) | 38.5 (32.2)
Statistical Analysis 1: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; p = 0.168, ANCOVA — [p-value comment as in outcome 3, analysis 1]

10. Secondary Outcome: Maximum Concentration (Cmax) of Prasugrel's Inactive Metabolites, R-95913, R-106583, and R-119251
Description: as for outcome 2
Time Frame: Day 1, Day 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: nanogram per milliliter (ng/mL)
Arm/Group | Prasugrel Healthy Participants | Prasugrel Sickle Cell Disease
Number analyzed (Participants) | 13 | 12
nanogram per milliliter (ng/mL)
  10 mg SD (overall) for R-95913 | 30.2 [23.0 to 39.8] | 45.4 [34.3 to 60.1]
  7.5 mg MD for R-95913 (N=9, 8) | 33.4 [24.6 to 45.3] | 36.3 [26.3 to 50.2]
  5 mg MD for R-95913 (N=4, 4) | 18.4 [11.7 to 29.1] | 34.4 [21.8 to 54.4]
  10 mg SD (overall) for R-106583 | 68.5 [56.3 to 83.3] | 59.8 [49.0 to 73.0]
  7.5 mg MD for R-106583 (N=9, 8) | 56.8 [45.7 to 70.6] | 38.7 [30.8 to 48.7]
  5 mg MD for R-106583 (N=4, 4) | 38.7 [28.0 to 53.7] | 34.8 [25.1 to 48.2]
  10 mg SD (overall) for R-119251 | 24.9 [20.0 to 31.1] | 26.5 [21.1 to 33.2]
  7.5 mg MD for R-119251 (N=9, 8) | 15.5 [10.7 to 22.4] | 15.9 [12.2 to 20.7]
  5 mg MD for R-119251 (N=4, 4) | 20.3 [15.8 to 25.9] | 15.5 [10.7 to 22.4]
Statistical Analysis 1: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(Cmax) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 1.50, 90% CI 2-sided [1.01 to 2.22] — This is the estimated value for 10 mg SD (overall) for the R-95913 metabolite
Statistical Analysis 2: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(Cmax) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 1.09, 90% CI 2-sided [0.751 to 1.58] — This is the estimated value for 7.5 mg MD for the R-95913 metabolite
Statistical Analysis 3: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(Cmax) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 1.87, 90% CI 2-sided [1.09 to 3.20] — This is the estimated value for 5 mg MD for the R-95913 metabolite
Statistical Analysis 4: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(Cmax) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 0.873, 90% CI 2-sided [0.660 to 1.15] — This is the estimated value for 10 mg SD (overall) for the R-106583 metabolite
Statistical Analysis 5: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(Cmax) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 0.681, 90% CI 2-sided [0.524 to 0.886] — This is the estimated value for 7.5 mg MD for the R-106583 metabolite
Statistical Analysis 6: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(Cmax) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 0.898, 90% CI 2-sided [0.612 to 1.32] — This is the estimated value for 5 mg MD for the R-106583 metabolite
Statistical Analysis 7: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(Cmax) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 1.06, 90% CI 2-sided [0.773 to 1.46] — This is the estimated value for 10 mg SD (overall) for the R-119251 metabolite
Statistical Analysis 8: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(Cmax) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 0.785, 90% CI 2-sided [0.582 to 1.06] — This is the estimated value for 7.5 mg MD for the R-119251 metabolite
Statistical Analysis 9: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; Mixed Models Analysis; Log(Cmax) = Participant + Population + Dose + Population*Dose + Random Error; Ratio of Geometric LS Means, SCD:Healthy = 1.00, 90% CI 2-sided [0.648 to 1.55] — This is the estimated value for 5 mg MD for the R-119251 metabolite

11. Secondary Outcome: Change From Baseline in the P2Y12 Reaction Units (PRU) Device Reported P2Y12 Percent Inhibition at Day 12
Description: PRU device reported VerifyNow percent inhibition is reported by Accumetrics VerifyNow™ P2Y12 (VN-P2Y12) assay, a point-of-care device that measures platelet aggregation with single-use, disposable cartridges.
Time Frame: Baseline, Day 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent inhibition
Arm/Group | Prasugrel Healthy Participants | Prasugrel Sickle Cell Disease
Number analyzed (Participants) | 11 | 11
percent inhibition
  Baseline (Day 1) | 12.0 (11.0) | 1.0 (2.2)
  Change from Baseline at Day 12 (N=11, 10) | 60.1 (19.6) | 47.9 (17.0)
Statistical Analysis 1: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; p = 0.060, ANCOVA — [p-value comment as in outcome 3, analysis 1]

12. Secondary Outcome: Change From Baseline in the Platelet Reactivity Index (PRI) of Prasugrel at Day 12
Description: PRI was calculated by vasodilator-associated phosphoprotein (VASP) phosphorylation assay using flow cytometry (FC) and a VASP assay using enzyme-linked immunosorbent assay (ELISA). The PRI indicates the level of P2Y12 inhibition. A low PRI reflects strong inhibition of P2Y12, whereas a high PRI reflects weak/absent inhibition of P2Y12.
Time Frame: Baseline, Day 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage PRI
Arm/Group | Prasugrel Healthy Participants | Prasugrel Sickle Cell Disease
Number analyzed (Participants) | 13 | 13
percentage PRI
  Flow Cytometry at Baseline (Day 1), (N=12, 8) | 78.91 (10.03) | 59.36 (23.31)
  Flow Cytometry, Day 12 Change, (N=12, 8) | -49.883 (22.004) | -46.000 (27.395)
  ELISA at Baseline (Day 1), (N=11, 13) | 94.70 (2.39) | 92.03 (5.65)
  ELISA, Day 12 Change (N=11, 12) | -70.436 (17.160) | -68.117 (12.856)
Statistical Analysis 1: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; p = 0.086, ANCOVA — This is the p-value for PRI by flow cytometry. The p-value is from model: Change from Baseline = Baseline + Treatment + Population + Treatment*Population + Random Error
Statistical Analysis 2: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; p = 0.679, ANCOVA — This is the p-value for PRI by ELISA. The p-value is from model: Change from Baseline = Baseline + Treatment + Population + Treatment*Population + Random Error

13. Secondary Outcome: Change From Baseline in the Area Under the Aggregation Curve at Day 12
Description: AUC to 20 micromolar (μM) adenosine diphosphate (ADP), 6.5μM ADP, Collagen, and thrombin receptor activator for peptide 6 (TRAP-6) were calculated by whole blood multi-electrode aggregometry (MEA) assay. Platelet aggregation was continuously recorded for 5 minutes and quantified as area under the aggregation curve, measured in aggregation units*minutes (AU*min).
Time Frame: Baseline, Day 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: aggregation units*minutes (AU*min)
Arm/Group | Prasugrel Healthy Participants | Prasugrel Sickle Cell Disease
Number analyzed (Participants) | 13 | 12
aggregation units*minutes (AU*min)
  AU*min to 6.5 µM ADP at Baseline (Day 1) | 76.5 (13.2) | 106.4 (27.9)
  AU*min to 6.5 µM ADP, Day 12 Change (N=13, 11) | -49.538 (17.145) | -63.182 (24.153)
  AU*min to 20 µM ADP at Baseline (Day 1) | 85.0 (19.0) | 108.1 (27.7)
  AU*min to 20 µM ADP, Day 12 Change (N=13, 11) | -54.077 (22.552) | -66.182 (26.084)
  AU*min to Collagen at Baseline (Day 1) | 85.5 (12.7) | 102.3 (25.4)
  AU*min to Collagen, Day 12 Change (N=13, 11) | -7.692 (11.707) | -3.000 (26.038)
  AU*min to TRAP-6 at Baseline (Day 1) | 120.2 (18.6) | 131.5 (30.7)
  AU*min to TRAP-6, Day 12 Change (N=13, 11) | -7.846 (20.136) | -2.818 (33.045)
Statistical Analysis 1: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; p = 0.396, ANCOVA — This is the p-value for AU*min to 6.5 µM ADP. The p-value is from model: Change from Baseline = Baseline + Treatment + Population + Treatment*Population + Random Error
Statistical Analysis 2: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; p = 0.288, ANCOVA — This is the p-value for AU*min to 20 µM ADP. The p-value is from model: Change from Baseline = Baseline + Treatment + Population + Treatment*Population + Random Error
Statistical Analysis 3: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; p = 0.095, ANCOVA — This is the p-value for AU*min to Collagen. The p-value is from model: Change from Baseline = Baseline + Treatment + Population + Treatment*Population + Random Error
Statistical Analysis 4: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; p = 0.086, ANCOVA — This is the p-value for AU*min to TRAP-6. The p-value is from model: Change from Baseline = Baseline + Treatment + Population + Treatment*Population + Random Error

14. Secondary Outcome: Change From Baseline in the Percent Aggregation to 20 µM Adenosine Diphosphate (ADP) at Day 12
Description: Percent aggregation was assessed by Plateletworks® ADP assay, a whole blood-based test of platelet aggregation for the assessment of platelet inhibition. The assay determines the change in single platelet count due to activation and aggregation by ADP and inhibition thereof by antiplatelet agents.
Time Frame: Baseline, Day 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent aggregation
Arm/Group | Prasugrel Healthy Participants | Prasugrel Sickle Cell Disease
Number analyzed (Participants) | 13 | 12
percent aggregation
  Baseline (Day 1) | 91.3 (9.8) | 74.0 (30.0)
  Change from Baseline at Day 12 (N=12, 10) | -53.0 (16.4) | -46.7 (44.8)
Statistical Analysis 1: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; p = 0.083, ANCOVA — [p-value comment as in outcome 3, analysis 1]

15. Secondary Outcome: P2Y12 Reaction Units (PRU)-Derived VerifyNow (VN) Percent Inhibition at Day 12
Description: PRU-derived VN percent inhibition is calculated as a percent decrease of PRU from baseline using the following formula:
  ([PRU at baseline - PRU at time of post baseline] / PRU at baseline) x 100%
Time Frame: Day 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent inhibition
Arm/Group | Prasugrel Healthy Participants | Prasugrel Sickle Cell Disease
Number analyzed (Participants) | 11 | 10
percent inhibition | 65.8 (23.4) | 47.8 (18.6)
Statistical Analysis 1: Comparison: Prasugrel Healthy Participants vs Prasugrel Sickle Cell Disease; Test type: Superiority or Other; p = 0.124, ANCOVA — [p-value comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Groups:
- Prasugrel 10/5 mg Healthy Participants: Participants received a single 10-milligram (mg) dose on Day 1 (single dose [SD]), followed by 5 mg/day (for participants<60 kilograms [kg]) for an additional 11 days (multiple dose [MD]).
- Prasugrel 10/7.5 mg Healthy Participants; Prasugrel 10/7.5 mg Sickle Cell Disease: Participants received a single 10-mg dose on Day 1 (SD), followed by 7.5 mg/day (for participants≥60 kg) for an additional 11 days (MD).
- All Prasugrel Healthy Participants; All Prasugrel Sickle Cell Disease Participants: Participants received a single 10-mg dose on Day 1 (SD), followed by either 5 mg/day (for participants<60 kg) or 7.5 mg/day (for participants≥60 kg) for an additional 11 days (MD).
- Prasugrel 10/5 mg Sickle Cell Disease: Participants received a single 10-mg dose on Day 1 (SD), followed by 5 mg/day (for participants<60 kg) for an additional 11 days (MD).
Arm/Group | Prasugrel 10/5 mg Healthy Participants | Prasugrel 10/7.5 mg Healthy Participants | All Prasugrel Healthy Participants | Prasugrel 10/5 mg Sickle Cell Disease | Prasugrel 10/7.5 mg Sickle Cell Disease | All Prasugrel Sickle Cell Disease Participants
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/9 | 0/13 | 0/4 | 0/9 | 0/13
Other Adverse Events (participants affected / at risk) | 3/4 | 5/9 | 8/13 | 3/4 | 7/9 | 10/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel 10/5 mg Healthy Participants (N=4) | Prasugrel 10/7.5 mg Healthy Participants (N=9) | All Prasugrel Healthy Participants (N=13) | Prasugrel 10/5 mg Sickle Cell Disease (N=4) | Prasugrel 10/7.5 mg Sickle Cell Disease (N=9) | All Prasugrel Sickle Cell Disease Participants (N=13)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ulcer (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 3 (5) | 6 (8) | 3 (3) | 4 (7) | 7 (10)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days